CLINICAL TRIAL: NCT07266987
Title: The Effect of Watching an Educational Video on Pain, Anxiety, and Comfort Levels in Patients Undergoing Thyroid Biopsy
Brief Title: Video Education and Patient Comfort in Thyroid Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: muş alpa
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Pain
Keywords: pain; patient; nursing care
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In the intervention group, patients will watch a short therapeutic and relaxing video immediately before and during the thyroid biopsy procedure. The video will be projected onto the wall in the interventional radiology room. The aim is to help patients relax, reduce anxiety, and improve comfort during the procedure. The control group will receive standard care without video intervention.
Who Masked: Outcomes Assessor
Masking Description: The data analyst was blinded to group allocation during the statistical analysis to prevent potential bias. Participant data were coded numerically, and the analyst did not have access to information identifying which participants belonged to the intervention or control group until the analysis was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Other: MULTİSENSORY Video
- Control Group (No Intervention)

INTERVENTIONS:
Other: MULTİSENSORY Video — The multisensory video is a short therapeutic and relaxing video designed to stimulate multiple senses-sight and hearing-simultaneously. It includes calming nature scenes, soft background music, and soothing narration to create a relaxing environment. The purpose of the multisensory video is to reduce anxiety, distract attention from the invasive procedure, and enhance patient comfort during the thyroid biopsy.
  Arms: experimental group

SUMMARY:
This quasi-experimental study aims to determine the effect of watching an educational and therapeutic video on patients' pain, anxiety, and comfort levels during thyroid biopsy procedures. The study will be conducted in the interventional radiology unit of Muş State Hospital between July 30, 2025, and August 28, 2026. A total of 68 patients (34 experimental and 34 control) will be included. Data will be collected using the Descriptive Information Form, Visual Analog Scale for Pain (VAS-Pain), State Anxiety Inventory, and Visual Analog Scale for Comfort (VAS-Comfort). The intervention group will watch a relaxing educational video immediately before and during the biopsy procedure, while the control group will receive standard care. Pre- and post-test measurements will be compared to evaluate changes in pain, anxiety, and comfort levels

DETAILED DESCRIPTION:
This research was designed as a quasi-experimental study with pretest and posttest measurements, based on epidemiological intervention methods. The study will take place in the interventional radiology unit of Muş State Hospital. The study population will include all patients who are admitted to the radiology unit for thyroid (goiter) biopsy. The sample size was calculated using the G*Power 3.1.9.7 program with a medium effect size (0.5), α=0.05, and power (1-β)=0.80, resulting in a total of 68 participants-34 in the intervention group and 34 in the control group.

Inclusion criteria: being literate and not having any psychiatric disorder. Exclusion criteria: having a psychological disorder that may affect the reliability of responses (e.g., bipolar disorder, dementia) or having undergone a thyroid biopsy before.

Participants will be assigned alternately: patients with odd numbers will be in the control group, and even numbers in the experimental group. The experimental group will watch a therapeutic (relaxing) video projected on the wall immediately before and during the biopsy. The video aims to reduce anxiety and discomfort associated with the procedure. Control group patients will receive the routine procedure without any additional intervention.

Data collection tools will include:

Descriptive Information Form: Prepared by researchers to record demographic and clinical characteristics.

Visual Analog Scale for Pain (VAS-Pain): Developed by Freyd (1983) to measure pain intensity on a 10-cm scale (0 = no pain, 10 = worst pain).

State Anxiety Inventory: Developed by Spielberger et al. (1970), validated in Turkish by Öner and Le Compte (1998), used to assess situational anxiety.

Visual Analog Scale for Comfort (VAS-Comfort): A 10-cm visual scale to evaluate patient comfort levels during the procedure (0 = least comfort, 10 = greatest comfort).

ELIGIBILITY:
Inclusion Criteria:

* Literate individuals who can read and write

Aged 18 years and older

Scheduled to undergo a thyroid (goiter) biopsy in the interventional radiology unit

Voluntarily agreeing to participate in the study and providing informed consent

Having no psychiatric diagnosis or cognitive impairment that may affect participation

Exclusion Criteria:

* Having a diagnosed psychological or psychiatric disorder that may affect response reliability (e.g., bipolar disorder, dementia, schizophrenia)

Having undergone a thyroid biopsy previously

Having visual or hearing impairments that prevent watching or understanding the video

Refusing to participate or withdrawing consent during the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The patient's pain level | 5 month
  Visual Analog Scale for Pain (VAS-Pain): Developed by Freyd (1983) to measure pain intensity on a 10-cm scale (0 = no pain, 10 = worst pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Muş State Hospital, Muş, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 1 years
Access Criteria: All information will be shared once it is provided.